CLINICAL TRIAL: NCT05231057
Title: Impact of Clinical Pilates Exercise on Pain, Cardiorespiratory Fitness, Functional Ability, And Quality of Life in Children With Polyarticular Juvenile Idiopathic Arthritis
Brief Title: Impact of Pilates Exercise in Children With Juvenile Idiopathic Arthritis
Acronym: Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qassim University (Other)
Collaborators: Cairo University (Other); Prince Sattam Bin Abdulaziz University (Other)
Responsible Party: Principal Investigator, Maged Basha, Assistant Professor, College of Medical Rehabilitation, Qassim University, Saudi Arabia, Qassim, Buraidah. Consultant Physical Therapist, El-Sahel Teaching Hospital, General Organization for Teaching Hospitals and Institutes, Cairo, Egypt., Qassim University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RHPT/0020/0035
Record Dates: First submitted 2022-01-28; First posted 2022-02-09 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Juvenile Arthritis; Cardiorespiratory Fitness; Quality of Life
MeSH Terms: conditions — Arthritis, Juvenile | interventions — Exercise Movement Techniques

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Patients in the study group received Pilates exercises plus conventional physical therapy program
  Interventions: Other: Pilates exercises; Other: Conventional physical therapy program
- control group (Experimental): Patients in the control group received conventional physical therapy
  Interventions: Other: Conventional physical therapy program

INTERVENTIONS:
Other: Pilates exercises — Mat, Pilates band or elastic bands, and Pilate's ball
  Other Names: Pilates band
  Arms: experimental group
Other: Conventional physical therapy program — pain relief, increasing flexibility, and mobility, improving muscle strength
  Other Names: pain reliving modalities, stretching exercises

SUMMARY:
Juvenile idiopathic arthritis (JIA) is one of the most common chronic childhood inflammatory diseases that is characterized by permanent joint inflammation attributable to immune system disturbance.

DETAILED DESCRIPTION:
Therapeutic exercises play an essential role as a non-pharmacologic treatment for children with JIA. It has effectively been used to reduce pain, improve muscular function, increase physical activity and promote quality of life in children with chronic musculoskeletal disorders. Clinical Pilates exercise is usually perceived as enjoyable activity by children with JIA, thereby, it can help them be more active for extended periods without causing discomfort while also allowing them to control their breathing and avoid becoming fatigued.

ELIGIBILITY:
Inclusion Criteria:

* Polyarticular JIA per the International League of Associations for Rheumatology classification.
* Age ranges from 10 to14 years.
* Stable medical treatment.

Exclusion Criteria:

* If they had contractures.
* Congenital anomalies.
* History of surgery.
* History of systemic disease
* Cardiorespiratory co-morbidity.
* Participation in regular exercises or sports activity.

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-07-25 (Actual); Study Completion 2021-12-05 (Actual)

PRIMARY OUTCOMES:
Pain assessment | at baseline
  measured using visual analog scale. A score of zero means no pain, while a score often means significant pain.
Pain assessment | after 12 weeks
  measured using visual analog scale. A score of zero means no pain, while a score often means significant pain.
Cardiorespiratory fitness assessment | at baseline
  assessed using electromagnetic cycle ergometer with electronic braking
Cardiorespiratory fitness assessment | after 12 weeks
  assessed using electromagnetic cycle ergometer with electronic braking

SECONDARY OUTCOMES:
Functional ability assessment | at baseline
  assessed using The Childhood Health Assessment Questionnaire
Functional ability assessment | after 12 weeks
  assessed using The Childhood Health Assessment Questionnaire
health-related quality of life | at baseline
  assessed using The self-report Pediatric Quality of Life Inventory
health-related quality of life | after 12 weeks
  assessed using The self-report Pediatric Quality of Life Inventory

CONTACTS AND LOCATIONS:
Overall Officials: Alshimaa Azab, PhD, Study Chair — Cairo University; Maged Basha, PhD, Study Director — Qassim University
Locations (1):
- Outpatient Clinic of College of Applied Medical Sciences, Prince Sattam bin Abdulaziz University, Al Kharj, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
The data sets generated during and/or analyzed during the current study are available from the corresponding author on reasonable request.
Supporting Information: Study Protocol
Time Frame: 6 months after publication
Access Criteria: relevance to the topic of the study and approval of all co-authors within 1 month of receiving the request.

REFERENCES:
- [Background] Franco CB, Ribeiro AF, Morcillo AM, Zambon MP, Almeida MB, Rozov T. Air stacking: effects of Pilates mat exercises on muscle strength and on pulmonary function in patients with cystic fibrosis. J Bras Pneumol. 2014 Oct;40(5):521-7. doi: 10.1590/s1806-37132014000500008. PMID 25410840
- [Result] Oen K, Duffy CM, Tse SM, Ramsey S, Ellsworth J, Chedeville G, Chetaille AL, Saint-Cyr C, Cabral DA, Spiegel LR, Schneider R, Lang B, Huber AM, Dancey P, Silverman E, Rosenberg AM, Cameron B, Johnson N, Dorval J, Scuccimarri R, Campillo S, Petty RE, Duffy KN, Boire G, Haddad E, Houghton K, Laxer R, Turvey SE, Miettunen P, Gross K, Guzman J, Benseler S, Feldman BM, Espinosa V, Yeung RS, Tucker L. Early outcomes and improvement of patients with juvenile idiopathic arthritis enrolled in a Canadian multicenter inception cohort. Arthritis Care Res (Hoboken). 2010 Apr;62(4):527-36. doi: 10.1002/acr.20044. PMID 20391508
- [Result] Haverman L, Grootenhuis MA, van den Berg JM, van Veenendaal M, Dolman KM, Swart JF, Kuijpers TW, van Rossum MA. Predictors of health-related quality of life in children and adolescents with juvenile idiopathic arthritis: results from a Web-based survey. Arthritis Care Res (Hoboken). 2012 May;64(5):694-703. doi: 10.1002/acr.21609. PMID 22238240